CLINICAL TRIAL: NCT04326894
Title: Methorexate and Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Anna Abou-Raya, MD, University of Alexandria
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: alexmed1391963211966
Record Dates: First submitted 2013-08-08; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Pain Reduction; Physical Function Improvement
Keywords: methotrxate, knee osteoarthritis, inflammation, pain, function
MeSH Terms: conditions — Osteoarthritis, Knee; Inflammation; Pain | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methotrexate (Experimental): 25mg oral MTX tablets
  Interventions: Drug: 25 mg/week oral methotrexate tablets
- Placebo (Placebo Comparator): 25 mg/week placebo tablets
  Interventions: Drug: 25mg/week oral placebo tablets

INTERVENTIONS:
Drug: 25 mg/week oral methotrexate tablets
  Other Names: interventional drug
  Arms: Methotrexate
Drug: 25mg/week oral placebo tablets
  Arms: Placebo

SUMMARY:
Osteoarthritis (OA) is considered a complex, multifactorial disease leading to considerable pain and functional disability amongst older adults in particular.Synovial inflammation and proliferation has emerged as a key component of OA and as a potential predictor of worsening disease. Methotrexate (MTX) is widely used in the treatment of all inflammatory rheumatic diseases. Accordingly, the aim of the present study is to assess the efficacy of methotrexate (MTX) in decreasing pain and inflammation in symptomatic knee OA.

128 patients with clinical and radiographic criteria of primary knee OA pain,were recruited. Patients meeting the eligibility criteria are randomized in a 1:1 ratio to receive either 25mg/week oral MTX (n=64) or placebo (n=64) together with their usual therapy provided the dosages are kept constant for 32 weeks. The primary outcome measure is pain reduction and secondary outcome measures is improvement in physical function scores.

Keywords:

methotrexate knee osteoarthritis inflammation pain reduction physical funtion

ELIGIBILITY:
Inclusion Criteria:

* primary knee osteoarthritis
* synovitis
* pain

Exclusion Criteria:

* other inflammatory conditions
* hepatic insufficiency
* renal insufficiency

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pain reduction | 8 months
  The primary outcome measure was pain reduction.Pain was assessed using the Visual Analogue pain Scale, (VAS, 0-100 mm).

SECONDARY OUTCOMES:
Physical function improvement | 8 months
  Functional assessment was performed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and Activities of daily living (ADL) scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Alexandria, Egypt